CLINICAL TRIAL: NCT06148090
Title: Screening for Adrenal Insufficiency During Dermocorticoid Reduction in Bullous Pemphigoid
Brief Title: Screening for Adrenal Insufficiency During Dermocorticoid Reduction in Bullous Pemphigoid (BP)
Acronym: PB-DEPIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2023/07
Record Dates: First submitted 2023-11-17; First posted 2023-11-28 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pemphigoid, Bullous; Adrenal Insufficiency
Keywords: Adrenal insufficiency; Iatrogenic; Bullous Pemphigoid; Topical corticosteroids
MeSH Terms: conditions — Pemphigoid, Bullous; Adrenal Insufficiency

STUDY DESIGN:
Intervention Model Description: At two occasions during the clobetasol decreasing, cortisol and ionogram measurement at 8 AM and clinical assessment by a physician:
  * Visit 1: 20-40 g clobetasol twice a week for at least 1 month
  * Visit 2: 20-40 g clobetasol once a week for at least 1 month A third visit (visit 3) is necessary if blood cortisol is between 138 and 500 nmol/L, to make a Synacthen® test (new cortisol dosage at 8 AM, then IM or IV injection of a 250 microgram ampoule of Synacthen® completed by a 2nd cortisol dosage one hour later)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated with clobetasol propionate (Experimental)
  Interventions: Diagnostic Test: clobetasol decreasing measurement

INTERVENTIONS:
Diagnostic Test: clobetasol decreasing measurement — At two occasions during the clobetasol decreasing measurement at 8 AM and clinical assessment by a physician:
  * Visit 1: 20-40 g clobetasol twice a week for at least 1 month
  * Visit 2: 20-40 g clobetasol once a week for at least 1 month

SUMMARY:
The braking of the corticotropic axis is well established during the induction phase of superpotent topical corticosteroid therapy (clobetasol propionate) in bullous pemphigoid (BP). But the evolution of the corticotropic axis in the following months, especially during the tapering of topical steroids has never been studied. The objective of this study is to evaluate the prevalence of adrenal insufficiency during the topical corticosteroid therapy tapering in patients treated according to current recommendations.

The secondary objectives of the study are :

* to evaluate the presence of other clinico-biological signs of adrenal insufficiency (hypotension, hypoglycemia and/or hyponatremia)
* to compare the characteristics of patients with adrenal insufficiency to those without in order to identify potential risk factors for adrenal insufficiency in BP.

DETAILED DESCRIPTION:
BP is the most common autoimmune bullous dermatosis, with 400 incident cases per year in France and an estimated annual mortality rate of 30%. It affects very old and frail patients, with an average age of 80 years.

High potency topical corticosteroids is the first line therapy, with a high dose applied to the entire tegument for at least 4 months according to current guidelines. In this high potency topical therapy, a braking of the corticotropic axis has been reported during the initial phase of treatment, at the highest doses, explained by the transdermal and systemic passage of dermocorticoids. Monitoring if natural cortisol secretion will start again has never been studied during the tapering of topical corticosteroid therapy, and its under-diagnosis could be deleterious for patients. The French guidelines currently recommends hydrocortisone supplementation at the time of waning from less than 20 g of clobetasol propionate per week, but without any data supporting it.

Prospective multicenter study coordinated by the Bordeaux Dermatology Department and conducted within the French study Group on autoimmune bullous diseases, will aim to include 50 patients with a diagnosis of bullous pemphigoid and treated according to recommendations.

Serum dosage of Cortisol concentration will be measured on two occasions, at the last two steps of the corticosteroid tapering (20-40g, twice a week and 20-40g once a week). If necessary, a Synacthen® test will be performed in addition.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age
* BP diagnosis with at least 3 of the following 4 criteria:

  * Age greater than 70 years
  * Absence of mucosal involvement
  * Absence of atrophic scarring
  * No predominance of head and neck
* Skin biopsy with subepidermal cleavage and :

  * FD with Ig and/or C3 deposits along the basement membrane
  * And/or positive serum anti-BP180 and/or anti-BP230 antibodies
* Treated with clobetasol propionate, with or without background treatment (methotrexate, mycophenolate mofetil, IV Ig, omalizumab, rituximab)
* Treatment with clobetasol propionate 0.05%, 20 to 40 g per application, twice a week for at least one month
* Affiliated to a social security regimen ( without AME)
* Free, informed and expressed consent (confirmed in writing)

Exclusion Criteria:

* Old or ongoing adrenal insufficiency
* Systemic corticosteroid therapy of more than 1 month in the previous 3 months and/or more than 3 months in the previous 12 months, or in the 7 days prior to the cortisol test
* Immuno-induced bullous pemphigoid (anti-PD1, PDL1 and/or anti-CTLA4)
* Impossible to perform a blood test between 7:30 and 8:30 am

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Measure of cortisol concentration in serum | Month 1
  Cortisol concentration in serum, after at least 1 month treatment with 20-40g of clobetasol twice a week
Measure of cortisol concentration in serum | Month 2
  Cortisol concentration in serum, after at least 1 month treatment with 20-40g of clobetasol one a week
Measure of cortisol concentration in serum after Adreno CorticoTropic Hormone (ACTH) stimulation test (Synacthen®) | Month 1
  ACTH stimulation test is necessary if serum cortisol concentration is found between 138 and 500 nmol/L
Measure of cortisol concentration in serum after ACTH stimulation test (Synacthen®) | Month 2
  ACTH stimulation test is necessary if serum cortisol concentration is found between 138 and 500 nmol/L

SECONDARY OUTCOMES:
Measure of glucose concentration in blood | Month 1
  Searching for a biological sign of adrenal insufficiency : hypoglycemia
Measure of glucose concentration in blood | Month 2
  Searching for a biological sign of adrenal insufficiency : hypoglycemia
Measure of sodium concentration in blood | Month 1
  Searching for a biological sign of adrenal insufficiency : hyponatremia
Measure of sodium concentration in blood | Month 2
  Searching for a biological sign of adrenal insufficiency : hyponatremia
Measure of blood pressure | Month 1
  Searching for a clinical sign of adrenal insufficiency : low blood pressure
Measure of blood pressure | Month 2
  Searching for a clinical sign of adrenal insufficiency : low blood pressure
Evaluation of skin atrophy (actinic purpura, skin thinness, post-blister erosion) | Month 1
  Evaluation of skin, looking for factors increasing clobetasol absorption and/or predicting adrenal insufficiency
Evaluation of skin atrophy (actinic purpura, skin thinness, post-blister erosion) | Month 2
  Evaluation of skin, looking for factors increasing clobetasol absorption and/or predicting adrenal insufficiency
Measure of Weight | Month 1
  Evaluating if low body mass index increases clobetasol absorption and/or predicts adrenal insufficiency
Measure of Weight | Month 2
  Evaluating if low body mass index increases clobetasol absorption and/or predicts adrenal insufficiency
Measure of Height | Month 1
  Evaluating if low body mass index increases clobetasol absorption and/or predicts adrenal insufficiency
Measure of Height | Month 2
  Evaluating if low body mass index increases clobetasol absorption and/or predicts adrenal insufficiency
Measure of Quantity of clobetasol applied per week | Month 1
  Evaluating if the risk of adrenal insufficiency depends of the quantity and/or duration of clobetasol treatment
Measure of Quantity of clobetasol applied per week | Month 2
  Evaluating if the risk of adrenal insufficiency depends of the quantity and/or duration of clobetasol treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anne Pham-Ledard, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (5):
- France (5):
  - University Hospital of Bordeaux - Hospital Saint André, Bordeaux
  - CH de Libourne, Libourne
  - CHU de Limoges, Limoges
  - Hôpital Saint louis, Paris
  - CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No